CLINICAL TRIAL: NCT04953533
Title: Research on New Technologies for Diagnosis and Treatment of Skin Diseases and Venereal Diseases and Rheumatoid Diseases-- Research and Development of a New Technology for Detection of Abnormal Excretion of Intestinal Uric Acid Involved in the Incidence of Gout
Brief Title: Research and Development of a New Technology for Detection of Abnormal Excretion of Intestinal Uric Acid Involved in the Incidence of Gout
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020C03044
Record Dates: First submitted 2021-03-16; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-01

CONDITIONS: Gout; Hyperuricemia; Gut Microbiota; Uric Acid; Genetic Loci; Single Nucleotide Polymorphism; Feces
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — for specific SNP and intestinal microflora
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with gout: 1. age:year of 25~60;
  2. consistent with the 2015 ACR gout diagnostic criteria ,and serum uric acid >420umol/L;
  3. The patient are willing to take part in our study.
  Interventions: Other: no intervention
- patients with hyperuricemia: 1. age:year of 25~60;
  2. A medical record in our hospital showed that the person is healthy, without key disease;
  3. serum uric acid >420umol/L without gout flares.
  Interventions: Other: no intervention
- healthy controls: 1. age:year of 25~60;
  2. A medical record in our hospital showed that the person is healthy, without key disease;
  3. serum uric acid ≤420umol/L.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
To evaluate differences in specific SNPs and intestinal microflora between patients with gout and hyperuricemia and healthy controls.

DETAILED DESCRIPTION:
1. To evaluate differences in specific SNPs and intestinal microflora between patients with gout and hyperuricemia and healthy controls.
2. to measure the level of uric acid in feces.

ELIGIBILITY:
gout

Inclusion Criteria:

1. age:year of 25~60;
2. Be consistent with the 2015 American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) gout diagnostic criteria ,and serum uric acid >420 μmol/L;
3. The patient are willing to take part in our study.

Exclusion Criteria:

1. abronia, surgery, postoperative, dehydration within 2 weeks, acute or chronic infectious diseases, severe trauma, malnutrition, diabetes, malignant tumors;
2. diagnosed as cardiovascular and cerebrovascular diseases within 3 months;
3. heart failure (New York Heart Academy，grade IV);
4. hepatic insufficiency ( Alanine transaminase or Aspartate aminotransferase ≥3×upper limit)；
5. chronic kidney disease or abnormal renal function( serum creatinine ≥1.5×upper limit)；
6. excessive drinking；
7. The investigators considered the patients unsuitable for inclusion in this study.

hyperuricemia:

Inclusion Criteria:

1. age:year of 25~60;
2. A medical record in our hospital showed that the person is healthy, without key disease;
3. serum uric acid >420μmol/L without gout flares. Exclusion Criteria:Same as the group of gout.

healthy controls:

Inclusion Criteria:

age:year of 25~60; A medical record in our hospital showed that the person is healthy, without key disease; serum uric acid ≤420μmol/L. Exclusion Criteria:Same as the group of gout.

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: gout，hyperuricemia and healthy controls in our hospital.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-07-06 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
the difference of the specific Single Nucleotide Polymorphisms(SNPs) | 2021.1.6--2021.12.31
  We will test the specific SNPs that we have selected before, such as rs670, rs671, rs1014290 and so on. The SNPs will be tested by Taqman SNP assay and verified by sequencing.
intestinal flora | 2021.1.6--2022.12.31
  Feces will be collected in gout, hyperuricemia patients and healthy subjects. ofIntestinal flora will be tested and analysed. The detailed measurement is as follows: Firstly, the DNA of feces will be extracted according to the protocol of Fecal DNA Extraction Kit. Then, the concentration and purity of fecal DNA will be tested by spectrophotometer. Sequencing of the V3-V4 region of the 16S ribosomal RNA gene, building a library and then sequencing the qualified libraries by Illumina Platform(MiSeq). Using the QIIME、UCLUST、SILVA and Kyoto Encyclopedia of Genes and Genomes(KEGG) database to comparison and screen the intestinal bacterial with statistical significance. Operational taxonomic unit (OTU), α-diversity, β-diversity indices and so on of the fecal microbiota will be analyzed in patients with gout and hyperuricemia and normal control.
feces uric acid level | 2021.1.6--2.22.12.31
  Feces uric acid level will be tested by uric acid assay kit and we will analyze the differences of feces uric acid level in gout, hyperuricemia patients and healthy subjects.

SECONDARY OUTCOMES:
the incidence of gout in patients with hyperuricemia | 2021.12.31--2023.12.31
  follow-up the patients with hyperuricemia for at least one year, calculate the incidence of hyperuricemia patients develop to gout.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyong Liu, PHD, Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine; Lei Liu, PHD, Study Director — Second Affiliated Hospital of Zhejiang University School of Medicine; Peiyu Zhang, MFA, Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang university,; Mo Chen, PHD, Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine; Jundi Wang, bachelor, Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang university,; Shunjie Hu, bachelor, Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang university,
Locations (1):
- the second affliated hospital of Zhejiang university School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
For the time being, we decided not to share individual participant data with other researchers